CLINICAL TRIAL: NCT04203199
Title: H-coil TMS to Reduce Pain: A Pilot Study Evaluating Relative Efficacy of the H1 vs H7 Coil
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institution
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00062742
Record Dates: First submitted 2019-12-16; First posted 2019-12-18 (Actual); Results first posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2022-04

CONDITIONS: Healthy; Chronic Pain; Opioid Use; Pain, Chronic
Keywords: Transcranial Magnetic Stimulation; Brain Stimulation; Healthy controls; Treatment
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: The proposed study will employ a 1-visit cross sectional, double-blind, placebo-controlled design to parametrically evaluate two promising treatment strategies of rTMS using the H1 and H7-coil for dlPFC stimulation (Strategy 1) or mPFC stimulation (Strategy 2), respectively. Participants will be randomized to receive TMS to the dlPFC or mPFC (50% at each site). This will be done in a cohort of healthy control individuals recruited from the local Wake Forest University (WFU) community. Quantitative Sensory Testing (QST) and subjective pain ratings will be measured before and after the rTMS session.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- First H1 coil, then H7 coil (Experimental): There will be 1 screening and 2 TMS visits. The procedures will be identical for each TMS visit, except for the type of TMS delivered (H1 or H7 coil). Each participant will be assigned to both coils, with TMS type. Participants assigned to this arm will receive the H1 coil at TMS visit 1, H7 coil at TMS visit 2
  Interventions: Device: Real rTMS to the mPFC using H7 Coil; Device: Real rTMS to the dlPFC using H1 Coil
- First H7 coil, then H1 coil (Experimental): There will be 1 screening and 2 TMS visits. The procedures will be identical for each TMS visit, except for the type of TMS delivered (H1 or H7 coil). Each participant will be assigned to both coils, with TMS type. Participants assigned to this arm will receive the H7 coil at TMS visit 1, H1 coil at TMS visit 2.
  Interventions: Device: Real rTMS to the mPFC using H7 Coil; Device: Real rTMS to the dlPFC using H1 Coil

INTERVENTIONS:
Device: Real rTMS to the mPFC using H7 Coil — This will be delivered with the Brainsway H7 coil system; 1200 pulses with the H7 coil helmet. Blinded using active/sham operator cards.
Device: Real rTMS to the dlPFC using H1 Coil — This will be delivered with the Brainsway H1 coil system; 3000 pulses with the H1 coil helmet. Blinded using active/sham operator cards.

SUMMARY:
Chronic pain is a serious public health problem with estimates as high as nearly half of the adult population experiencing some form of pain that lasts for more than 6 months. Chronic use of opiates is a rapidly escalating crisis in the United States, with over 4.3 million Americans dependent on opiate analgesics, an escalating rate of opiate overdose deaths, and a resurgence of intravenous heroin use leading to total societal cost exceeding $55 billion. While opiates are effective at treating acute pain, tolerance to the analgesic effects develops quickly, leading to high abuse liability and dependence potential. Consequently, the development of a new, non-pharmacologic intervention to treat pain, such as repetitive transcranial magnetic stimulation (rTMS), which would provide analgesic benefit while also directly remodeling the neural circuitry responsible for cognitive control over opiate craving, would fill an increasingly urgent public health need.

DETAILED DESCRIPTION:
Chronic pain is a serious public health problem with estimates as high as nearly half of the adult population experiencing some form of pain that lasts for more than 6 months. Chronic use of opiates is a rapidly escalating crisis in the United States, with over 4.3 million Americans dependent on opiate analgesics, an escalating rate of opiate overdose deaths, and a resurgence of intravenous heroin use leading to total societal cost exceeding $55 billion. While opiates are effective at treating acute pain, tolerance to the analgesic effects develops quickly, leading to high abuse liability and dependence potential. Consequently, the development of a new, non-pharmacologic intervention to treat pain, such as repetitive transcranial magnetic stimulation (rTMS), which would provide analgesic benefit while also directly remodeling the neural circuitry responsible for cognitive control over opiate craving, would fill an increasingly urgent public health need.

Acute pain is associated with elevated magnetic resonance imaging (MRI) blood-oxygen-level-dependent (BOLD) signal in targets of ascending nociceptive fibers including the insula, dorsal anterior cingulate (dACC), thalamus and somatosensory cortex - the 'Pain Network'. Perceived pain, and corresponding BOLD signal in the Pain Network, is attenuated by 10 Hz rTMS (a form of brain stimulation that results in long term potentiation (LTP) to the left dorsolateral prefrontal cortex (dlPFC, a node of the Executive Control Network). Dr. Borckardt was the first person to demonstrate that when LTP-like dlPFC rTMS was delivered in the postoperative recovery room, patients used less morphine in the hospital and require less morphine long-term. These analgesic effects are now widely known, with over 33 clinical trials utilizing rTMS as a tool to decrease acute and chronic pain in various clinical populations.

These data all suggest that LTP-like DLPFC rTMS is a very strong candidate alleviating chronic pain (LTP-like dlPFC rTMS (Strategy 1, Aim 1)). An alternative approach, however, *which may also target opiate craving*, is to attenuate the Pain Network (through long term depression (LTD) of the ventromedial PFC) (LTD-like mPFC rTMS, Strategy 2, Aim 1). In a cohort of 49 individuals with chronic pain, Dr. Hanlon (Primary Investigator) recently demonstrated that LTD-like mPFC rTMS reduced baseline BOLD signal in multiple regions of interest (ROIs) *involved in craving which also overlap with the Pain Network* (e.g. dACC and Insula). To parametrically evaluate these 2 promising treatment strategies, the investigator has developed a 1-visit cross-sectional design wherein a cohort of healthy control individuals will receive Quantitative Sensory Testing before and after rTMS with the H1 and H7-coil for dlPFC stimulation (Strategy 1) and mPFC depression (Strategy 2), respectively. The investigator aims to:

Aim 1. Quantify the effects of LTP-like and LTD-like RTMS on Quantitative Sensory Testing Hypothesis: The pressure pain tolerance of individuals in these two groups will increase after one session of rTMS administered by the H1- and H7-coil design.

Aim 2. Evaluate the effects of rTMS on subjective experience of discomfort. Hypothesis: Subjective experience of discomfort will decrease in individuals after one session of LTP-like or LTD-like rTMS administered to the dlPFC and mPFC, respectively.

The relative efficacy of Strategy 1 vs 2 will directly translate to development of a large clinical trial of rTMS as an innovative, new treatment option for pain in opiate dependent individuals.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 65 (to maximize participation).
2. Does not have a history of and is currently not experiencing chronic pain.
3. Able to read and understand questionnaires and informed consent.
4. Lives within 50 miles of the study site.
5. Is not at elevated risk of seizure (i.e., does not have a history of seizures, is not currently prescribed medications known to lower seizure threshold).
6. Does not have a history of traumatic brain injury, including a head injury that resulted in hospitalization, loss of consciousness for more than 10 minutes, or having ever been informed that they have an epidural, subdural, or subarachnoid hemorrhage.

Exclusion Criteria:

1. Any psychoactive illicit substance use (except marijuana and nicotine) within the last 30 days by self-report and urine drug screen. For marijuana, no use within the last seven days by verbal report and negative (or decreasing) urine THC levels.
2. Meets DSM-V criteria for moderate substance dependence, current axis I disorders of major depression, panic disorder, obsessive-compulsive disorder, post traumatic stress syndrome, bipolar affective disorder, schizophrenia, dissociate disorders, eating disorders, and any other psychotic disorder.
3. Has current suicidal ideation or homicidal ideation.
4. Has the need for maintenance or acute treatment with any psychoactive medication including anti-seizure medications and medications for ADHD.
5. Females of childbearing potential who are pregnant (by urine HCG), nursing, or who are not using a reliable form of birth control.
6. Has current charges pending for a violent crime (not including DUI related offenses).
7. Suffers from chronic migraines.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2022-10-06 (Actual); Study Completion 2022-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Hanlon, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 8 screen failures. Only 31 randomized.
Period: First Intervention Period
Arm/Group | First H1 Coil, Then H7 Coil | First H7 Coil, Then H1 Coil
Started | 15 | 16
Completed | 15 | 15
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Period: Second Intervention Period
Arm/Group | First H1 Coil, Then H7 Coil | First H7 Coil, Then H1 Coil
Started | 15 | 15
Completed | 14 | 15
Not Completed | 1 | 0
Not completed — Medication change | 1 | 0

BASELINE CHARACTERISTICS:
Population: Includes subjects who randomized only.
Groups:
- Total: Total of all reporting groups
Arm/Group | First H1 Coil, Then H7 Coil | First H7 Coil, Then H1 Coil | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.27 (15.0) | 43.88 (15.4) | 47.45 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 3 | 5 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 13 | 14 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 15 | 16 | 31

OUTCOME MEASURES:

1. Primary Outcome: Changes in Painfulness Thresholds Using the Quantitative Pain Testing (QST) Task, Which Utilizes Pressure From the Medoc Algomed Device (Measured in kiloPascals).
Description: Based on pilot data, the investigators expect an interaction between treatment (DLPFC or MPFC TMS) and time (Before vs. After rTMS) on reported painfulness using a quantitative sensory testing technique which determines the sensation and pain thresholds of pressure. Painfulness ratings will be assessed and reported before and after rTMS.
Time Frame: rTMS treatment visit, an average of 2 and a half hours
Measure: Mean (Standard Deviation); unit: kPascals
Groups:
- Real rTMS to the mPFC Using H7 Coil: One session of low frequency repetitive transcranial magnetic stimulation (rTMS) will be delivered to the left medial prefrontal cortex (mPFC) using the H7-coil (20 min total, 1200 pulses delivered at 1 Hz continuously, 1 train, 120% resting motor threshold (rMT)). Real rTMS to the mPFC using H7 Coil: This will be delivered with the Brainsway H7 coil system; 1200 pulses with the H7 coil helmet. Blinded using active/sham operator cards.
- Real rTMS to the dlPFC Using H1 Coil: One session of high frequency repetitive transcranial magnetic stimulation (rTMS) will be delivered to the left dorsolateral prefrontal cortex (dlPFC) using the H1-coil (20 min total, 3000 pulses delivered at 10 Hz, 60 trains, 50 pulses/train, 5 sec on/15 sec off, 120% resting motor threshold (rMT)). Real rTMS to the dlPFC using H1 Coil: This will be delivered with the Brainsway H1 coil system; 3000 pulses with the H1 coil helmet. Blinded using active/sham operator cards.
Arm/Group | Real rTMS to the mPFC Using H7 Coil | Real rTMS to the dlPFC Using H1 Coil
Number analyzed (Participants) | 29 | 29
kPascals | 1.1 (101.3) | -23.4 (89)

2. Secondary Outcome: Changes in Pain Tolerance Thresholds Using the Quantitative Pain Testing (QST) Task, Which Utilizes Pressure From the Medoc Algomed Device (Measured in kiloPascals).
Description: The investigators do not expect an interaction between treatment (DLPFC or MPFC TMS) and time (Before vs. After rTMS) on pain tolerance thresholds using a quantitative sensory testing technique which determines the sensation and pain thresholds of pressure. Pain tolerance ratings will be assessed and reported before and after rTMS.
Time Frame: rTMS treatment visit, an average of 2 and a half hours
Measure: Mean (Standard Deviation); unit: kPascals
Arm/Group | Real rTMS to the mPFC Using H7 Coil | Real rTMS to the dlPFC Using H1 Coil
Number analyzed (Participants) | 29 | 29
kPascals | 4.8 (117.9) | 24.2 (134.4)

ADVERSE EVENTS:
Time Frame: Baseline through end of second visit - time frame varied. Two weeks maximum
Arm/Group | Real rTMS to the mPFC Using H7 Coil | Real rTMS to the dlPFC Using H1 Coil
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 0/29 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-14): https://cdn.clinicaltrials.gov/large-docs/99/NCT04203199/Prot_SAP_001.pdf
  • Informed Consent Form (2021-12-20): https://cdn.clinicaltrials.gov/large-docs/99/NCT04203199/ICF_000.pdf